CLINICAL TRIAL: NCT05427682
Title: A Single-center, Non-randomized, Open, Single-dose Clinical Trial to Evaluate the Pharmacokinetics and Safety of Pyroglutamate Rongliflozin Capsules in Subjects With Mild and Moderate Liver Damage
Brief Title: A Clinical Trial to Evaluate the Pharmacokinetics and Safety of Pyroglutamate Rongliflozin Capsules in Subjects With Mild and Moderate Liver Damage
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sunshine Lake Pharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DJT1116PG-DM-105
Record Dates: First submitted 2022-06-17; First posted 2022-06-22 (Actual); Last update posted 2022-06-22 (Actual); Status verified 2022-06

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group A (normal liver function) (Experimental): Each subject will receive a single dose of rongliflozin on Day 1
  Interventions: Drug: pyroglutamate rongliflozin capsules
- Group B (mild liver damage) (Experimental): Each subject will receive a single dose of rongliflozin on Day 1
  Interventions: Drug: pyroglutamate rongliflozin capsules
- Group C (normal liver function) (Experimental): Each subject will receive a single dose of rongliflozin on Day 1
  Interventions: Drug: pyroglutamate rongliflozin capsules
- Group D (moderate liver damage) (Experimental): Each subject will receive a single dose of rongliflozin on Day 1
  Interventions: Drug: pyroglutamate rongliflozin capsules

INTERVENTIONS:
Drug: pyroglutamate rongliflozin capsules — Subjects will receive one 50mg capsule on Day 1

SUMMARY:
To evaluate the pharmacokinetic characteristics of pyroglutamate rongliflozin capsules in subjects with mild and moderate liver damage and healthy subjects

ELIGIBILITY:
Inclusion Criteria:

* Sign the informed consent form before the experiment, understand and abide by the research process, and participate voluntarily;
* Adult subjects between the ages of 18 and 70 (including boundary values), both male and female;
* Female subjects or male subjects with potential fertility must agree to use effective contraceptive methods (see Appendix 2 for specific contraceptive methods) from signing informed consent to taking the trial drug within 4 weeks to avoid pregnancy or make their partners pregnant.
* The following selection criteria are only applicable to healthy subjects with normal liver function (groups A and C): the gender and age (+ or - 5 years) of subjects in groups A and C are matched with subjects in groups B and D respectively;
* The following selection criteria are only applicable to healthy subjects with normal liver function (groups A and C): body mass index (BMI): 18-30kg/m2 (including cut-off value) [BMI=weight (kg)/height 2 (m2) )] (BMI matching between groups A and C and groups B and D is + or - 15%);
* The following selection criteria are only applicable to healthy subjects with normal liver function (groups A and C): medical history, physical examination, vital signs monitoring, electrocardiogram, laboratory tests (blood routine, urine routine, blood biochemistry, coagulation) Function), alpha-fetoprotein (AFP), abdominal B-ultrasound (liver, spleen, gallbladder, pancreas, kidneys), and chest radiographs have normal or abnormal results, but the investigator judges them to be of no clinical significance.
* The following selection criteria are only applicable to subjects with liver dysfunction (groups B and D): for subjects with liver dysfunction without ascites, subclinical ascites, clinically mild and moderate ascites detected only by ultrasound or other imaging , Allow the body mass index (BMI) to be between 18-30 kg/m2 (including the critical value) [BMI= weight (kg) / height 2 (m2)];
* The following selection criteria are only applicable to subjects with liver dysfunction (groups B and D): according to the Child-Pugh classification (see Appendix 3) at the time of screening to evaluate the severity of patients with liver dysfunction in accordance with: (Grade A/Mild: Child -Pugh score 5 or 6 points; B grade/moderate: Child Pugh score 7-9 points);
* The following selection criteria are only applicable to subjects with liver dysfunction (groups B and D): combined with previous medical history, physical examination results, serological indicators (such as albumin, ALT, AST, bilirubin, prothrombin time, INR, etc.) ) And one of the following tests performed with standard diagnostic and treatment methods that meets the diagnostic basis for chronic liver disease: liver biopsy, computed tomography, magnetic resonance imaging, ultrasound, radioactive liver/spleen scan, laparoscopy;
* The following selection criteria are only applicable to subjects with liver damage (groups B and D): within 1 month before taking the test drug or 5 half-lives of the concomitant drug (whichever is longer) to the end of the study Those who have stable medication regimens for the treatment of liver dysfunction, liver disease complications and other concomitant diseases without adjustment (including the type of medication, dosage, or frequency of medication) or those who have not taken medication before enrollment; however, the study doctor's judgment does not affect Except for the adjustment of subject safety and pharmacokinetic endpoints;
* The following selection criteria are only applicable to subjects with liver dysfunction (groups B and D): the investigator judges that the liver function status of the subjects is stable and will not deteriorate significantly during the period from 1 month before taking the test drug to the end of the study By.

Exclusion Criteria:

* The subject has a history of severe allergies or allergies to the test drug and any of its components or related excipients;
* People with history of gastrointestinal or kidney disease or surgery (except for uncomplicated appendicitis resection and hernia repair) that may potentially affect the absorption, distribution, metabolism, and excretion of the test drug in the 6 months prior to screening, or the presence can make compliance People with reduced disease;
* The researcher judged that he currently has bleeding disorders, such as gastric and duodenal ulcers;
* People with a history of liver cancer or other malignant tumors before signing the informed consent form [exceptions: specific cancers (basal cell carcinoma of the skin, squamous cell carcinoma, or cervical carcinoma in situ, etc.) that are surgically removed and completely cured can be selected] or are currently assessed for existence People with potential malignant tumors;
* Patients with a history of repeated urinary tract infections or/and genital infections within 6 months before screening (recurrent urinary tract infection is defined as: repeated urinary tract infections > or = 2 times within 6 months, or repeated urinary tract infections in the past 12 months Infection > or =3 times);
* People with a history of recurring severe unconscious hypoglycemia (repeated severe hypoglycemia is defined as: 2 severe neurological symptoms in 4 weeks, hypoglycemia requiring the assistance of others to treat, or 2 blood glucose in 4 weeks< 3.0 mmol/L, or blood glucose < or = 3.9 mmol/L > or =3 times detected within 1 week);
* People with a history of alcoholism (alcoholism is defined as: drinking 14 units of alcohol per week: 1 unit = 285 mL of beer, or 25 mL of spirits, or 100 mL of wine) or those who have a positive alcohol breath test during the screening period;
* Those who have a history of drug abuse or have used drugs within 2 years before screening or those who have a positive urine drug screening during the screening period;
* Those who smoked more than 5 cigarettes a day in the 3 months before screening or who could not give up smoking from signing informed consent to leaving the group;
* Treponema pallidum antibody and/or human immunodeficiency virus (HIV) antibody test results are positive;
* Have taken food or drinks that affect CYP3A4 metabolic enzymes, such as grapefruit or drinks containing grapefruit within 7 days before the first medication;
* Consume chocolate, any food or drink that contains caffeine or is rich in xanthine within 72 hours before the first medication;
* Have taken any alcohol-containing products within 48 hours before the first medication;
* Those who donated blood > or = 400 mL or a large amount of blood loss within 3 months before screening, or who have a history of blood transfusion within 1 month before screening, or who plan to donate blood within 1 month after the end of the test;
* Have taken similar SGLT-2 inhibitor drugs within 14 days before screening or participated in other clinical trials within 3 months before screening (if the subject withdrew from the study before treatment, that is, not randomized or received treatment, they can be included in the group Research);
* The subject is breastfeeding or the result of serum pregnancy is positive;
* Take the prohibited concomitant medications within 1 month before taking the trial drug or within the 5 half-life period of the concomitant medication (whichever is the longer) to the end of the study (see Chapter 5.5.1 for details);
* The investigator believes that there are other subjects who are not suitable for participating in this trial (such as inability to tolerate oral drugs, poor peripheral venous access conditions, or significant risks to the subjects, etc.).
* The following exclusion criteria are only applicable to healthy subjects with normal liver function (groups A and C): hepatitis B surface antigen (HBsAg) and hepatitis C virus (HCV) antibody test results are positive;
* The following exclusion criteria are only applicable to healthy subjects with normal liver function (groups A and C): the subjects have the following clinically significant diseases before screening, including but not limited to gastrointestinal tract, kidney, liver, nerve, blood , Endocrine, tumor, lung, immune, mental or cardiovascular and cerebrovascular diseases;
* The following exclusion criteria are only applicable to healthy subjects with normal liver function (groups A and C): any prescription drugs, non-prescription drugs, any vitamin products or Chinese herbal medicines have been taken within 2 weeks before the first medication.
* The following exclusion criteria are only applicable to subjects with liver dysfunction (groups B and D): the laboratory test results at the time of screening meet any of the following: a) ALT>10×ULN; b) absolute value of neutrophils <0.75 ×109/L; c) platelets <50×109/L (except for cases in a stable state as judged by the investigator); d) hemoglobin <60 g/L; e) AFP>100 ng/mL; if 20 ng/ mL=AFP=100 ng/mL, liver ultrasonography or other imaging examinations (CT, MRI, etc.) are required to exclude subjects suspected of hepatocellular carcinoma; f) Estimated using the modified dietary test for kidney disease (MDRD) formula Glomerular filtration rate (eGFR) <60 mL/min/1.73m2 (for eGFR estimation formula, please refer to Appendix 4).
* The following exclusion criteria are only applicable to subjects with liver dysfunction (groups B and D): those with cardiovascular and cerebrovascular events within 6 months before screening, including stroke (except for lacunar infarction), acute myocardial infarction, cardiac Dysfunction (New York College of Cardiology [NYHA] Grade III or IV, see Appendix 6), transient ischemic attack, coronary intervention (including stent thrombosis), peripheral vascular intervention, unstable angina, etc.;
* The following exclusion criteria are only applicable to subjects with liver dysfunction (groups B and D): subjects who have severe esophageal and gastric varices or have undergone portal venous shunt, including transjugular intrahepatic portosystemic shunt Surgery (TIPS);
* The following exclusion criteria are only applicable to subjects with liver dysfunction (groups B and D): subjects suffering from biliary obstruction and other diseases that affect bile excretion or drug-induced liver injury;
* The following exclusion criteria are only applicable to subjects with liver damage (groups B and D): subjects suffering from liver failure or severe complications of liver cirrhosis (such as spontaneous bacterial peritonitis, bleeding from esophageal and gastric fundus veins, liver and kidney Syndrome, etc.);
* The following exclusion criteria are only applicable to subjects with liver damage (groups B and D): a history of liver transplantation;
* The following exclusion criteria are only applicable to subjects with liver damage (groups B and D): any prescription drugs, over-the-counter drugs, and any vitamins other than those used to treat liver damage or their comorbidities have been used within 2 weeks before the first medication Products or Chinese herbal medicine;
* The following exclusion criteria are only applicable to subjects with liver dysfunction (groups B and D): the investigator is based on the subject's medical history, physical examination, vital signs, laboratory tests (blood routine, urine routine, blood biochemistry, coagulation function) , AFP, 12-lead electrocardiogram, EEG, and judge that the subject has other clinically significant abnormalities (except for abnormal indexes related to liver function, HBsAg and HCV antibody positive), such as uncontrolled heart, breathing, gastrointestinal Tract, blood, nerve, or other diseases that may interfere with the subject's treatment, evaluation, or compliance with the research protocol, and those who are not suitable for inclusion in this study will also be excluded.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2022-04-19 (Actual); Primary Completion 2023-03-04 (Estimated); Study Completion 2023-06-02 (Estimated)

PRIMARY OUTCOMES:
Plasma concentrations of rongliflozin | 0 hour（pre-dose） to 96 hours after administration
  Plasma concentrations of rongliflizin following the administration of a single dose of rongliflozin, the pharmacokinetic parameters for rongliflozin will be measured in varying degrees of liver function.

SECONDARY OUTCOMES:
Incidence of Adverse Events [safety] | Day -1 (Baseline) to Day 5
  To evaluate the safety of pyroglutamate rongliflozin capsules in subjects with mild to moderate liver damage and healthy subjects

CONTACTS AND LOCATIONS:
Locations (1):
- West China Hospital of Sichuan University, Chengdu, Sichuan, China